CLINICAL TRIAL: NCT00388492
Title: BLADE: "A Comparison of Once Daily LPV/r to LPV/r BID in HIV-Infected Virologically Controlled Antiretroviral Experienced Subjects"
Brief Title: BLADE: Comparison of Once Daily Lopinavir/Ritonavir to Lopinavir/Ritonavir BID Dosing in HIV-Infected Subjects
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Bellos, Nicholaos C., M.D. (Individual)
Other Study IDs: 70-1002-075
Record Dates: First submitted 2006-10-12; First posted 2006-10-16 (Estimated); Last update posted 2007-01-11 (Estimated); Status verified 2006-10

CONDITIONS: HIV Infections
Keywords: HIV Infected
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The goal of this study is to evaluate the proportion of subjects both antiretroviral experienced and virologically suppressed on lopinavir/ritonavir (LPV/r)400/100mg twice daily who maintain viral suppression after switching to lopinavir/ritonavir (LPV/r)800/200mg once daily.

The hypothesis for this study is that the majority of subjects will remain virologically suppressed with once daily dosing versus twice daily dosing and therefore quality of life will be improved with the once daily dosing of lopinavir/ritonavir (LPV/r)800/200mg.

ELIGIBILITY:
Inclusion Criteria:

* Documentation HIV infection
* Male or Female
* 18 years of age
* Previously failed an NNRTI and/or 1 previous PI containing regimen
* Currently virologically controlled (VL<50 copies/mL) on a LPV/r containing regimen ≥ 3 months
* Any CD4+ cell count
* Cognitive ability to understand and provide written informed consent and willingness to participate in and comply with the study protocol
* Patient does not currently have or has not been treated for an active opportunistic infection (OI) consistent with CDC definition (Appendix B) within 30 days of screening
* Vital signs, physical examination and laboratory results do not exhibit evidence of acute illness
* A female is eligible to enter and participate in this study if she is of:

  * Non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal) or
  * Child-bearing potential, has a negative serum pregnancy test at screen, and agrees to one of the following:

    * Complete abstinence from intercourse from 2 weeks prior to administration of the study drug, throughout the study, and for at least 2 weeks after completion or premature discontinuation of the study to account for elimination of the investigational drug. Should a patient decide to become sexually active during the course of the study, she must be counseled and be willing to use one of the birth control methods below:
    * Double barrier method (male condom/spermicide, male condom/diaphragm, diaphragm/spermicide)
    * Any intrauterine device(IUD) with published data showing that the expected failure rate is <1% per year (not all IUD's meet this criterion)
    * Sterilization (female patient or male partner of female patient)
    * Any other methods with published data showing that the lowest expected failure rate for that method is <1% per year NOTE: Data are insufficient to exclude a clinically important interaction of LPV/r with drugs, such as hormonal contraceptives, that are highly metabolized by the cytochrome P450 enzyme system. As a result, hormonal contraception is not considered adequate.

Exclusion Criteria:

* Pregnancy or breastfeeding
* Hemodialysis or peritoneal dialysis
* Patients unable to provide written informed consent
* Use of concurrent medications known to affect lopinavir and/or ritonavir concentrations (as listed in the attached Kaletra package insert)
* Patient with active AIDS-defining opportunistic infection or disease according to the 1993 CDC AIDS surveillance definition (Clinical Category C) that, in the opinion of the investigator, would prelude the patient from participating in the study (See Appendix B)
* History of active substance abuse, excluding cannabis, or psychiatric illness that, in the opinion of the investigator, would preclude compliance with the protocol, dosing schedule and assessments.
* Patient is either pregnant at the time of screening evaluation or breast-feeding
* Patient, in the opinion of the investigator, is unlikely to be able to complete the 48-week dosing period and protocol evaluations and assessments or adhere to the study drug regimen
* Patient suffers from a serious medical condition, such as diabetes, congestive heart failure, cardiomyopathy or other cardiac dysfunction, which in the opinion of the investigator would compromise the safety of the patient
* Patient has malabsorption syndrome or other gastrointestinal dysfunction, which may interfere with drug absorption or render the patient unable to take oral medication
* HBV coinfection
* Patient has any of the following laboratory results within 30 days prior to the first dose of study medication:

  * Hemoglobin concentration <8.0g/dl
  * Absolute neutrophil count <750cells/mm3
  * Platelet count <50,000cells/mm3
  * Aminotransferase (AST, ALT) >3 times ULN
  * Serum creatinine >1.5 times the Upper Limits of Normal (ULN)
* Patient has required treatment with radiation therapy or cytotoxic chemotherapeutic agents within 4 weeks prior to entry, or has an anticipated need for these agents within the study period
* Patient requires treatment with immunomodulating agents, such as systemic corticosteroids, interleukins, or interferon's within 4 weeks prior to study entry, or patients who have received an HIV immunotherapeutic vaccine within 3 months prior to entry. Asthmatic patients using inhaled corticosteroids are eligible for enrollment.
* Patient receiving methadone therapy
* Patients requiring foscarnet therapy or therapy with other agents with documented activity against HIV-1 invitro
* Patient prescribed/taking astemizole, terfenadine, cisapride, midazolam, triazolam, flecainide, pimozide, propafenone, St. John's Wort, lovastatin, simvastatin, and rifampin or ergot derivatives (see section 5.5 Concomitant Medications and Non-Drug Therapies and Appendix C
* Patient has a history of allergy to any of the study drugs or any excipients therein.
* In addition, patients non-compliant with study medication during 2-4 week study periods despite adherence counseling will not be retained in the study due to increased risk for selective pressure and potential development of protease resistance.
* Patient requires inhaled or intranasal fluticasone

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 45

CONTACTS AND LOCATIONS:
Overall Officials: Nicholaos C. Bellos, MD, Principal Investigator — Nicholaos C. Bellos, MD
Locations (1):
- Nicholaos C. Bellos, MD, Dallas, Texas, United States